CLINICAL TRIAL: NCT04322682
Title: Colchicine Coronavirus SARS-CoV2 Trial (COLCORONA)
Acronym: COVID-19
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to several considerations (logistical, human and budgetary), the study was stopped early.
Sponsor: Montreal Heart Institute (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Bill and Melinda Gates Foundation (Other); The Government of Quebec (Other Government); Dacima Software Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MHIPS-2020-001; 3R01HL146206-02S1 (NIH)
Record Dates: First submitted 2020-03-23; First posted 2020-03-26 (Actual); Results first posted 2021-09-08 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-11

CONDITIONS: Corona Virus Infection
MeSH Terms: conditions — Coronavirus Infections | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: This will be a randomized, double-blind, placebo-controlled, multi-center study. Following signature of the informed consent form, approximately 6000 subjects meeting all inclusion and no exclusion criteria will be randomized to receive either colchicine or placebo (1:1 allocation ratio) for 30 days. Follow-up phone or video assessments will occur at 15 and 30 days following randomization for evaluation of the occurrence of any trial endpoints or other adverse events.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colchicine (Active Comparator): Patients will receive study medication colchicine 0.5 mg per os (PO) twice daily for the first 3 days and then once daily for the last 27 days. If a dose is missed, it should not be replaced.
  Interventions: Drug: Colchicine
- Placebo (Placebo Comparator): Patients will receive a placebo per os (PO) twice daily for the first 3 days and then once daily for the last 27 days. If a dose is missed, it should not be replaced.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Colchicine — Patients in this arm will receive study medication colchicine 0.5 mg per os (PO) twice daily for the first 3 days and then once daily for the last 27 days. If a dose is missed, it should not be replaced.
  Other Names: Immuno-modulatory
  Arms: Colchicine
Drug: Placebo oral tablet — Patients will receive the placebo 0.5 mg per os (PO) twice daily for the first 3 days and then once daily for the last 27 days. If a dose is missed, it should not be replaced.
  Arms: Placebo

SUMMARY:
This is a phase 3, randomized, double-blind, placebo-controlled multicenter study to evaluate the efficacy and safety of colchicine in adult patients diagnosed with COVID-19 infection and have at least one high-risk criterion. Approximately 6000 subjects meeting all inclusion and no exclusion criteria will be randomized to receive either colchicine or placebo tablets for 30 days.

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether short-term treatment with colchicine reduces the rate of death and lung complications related to COVID-19. The secondary objective is to determine the safety of treatment with colchicine in this patient population.

Approximately 6000 patients will be enrolled to receive either colchicine or placebo (1:1 allocation ratio) for 30 days. Follow-up assessments will occur at 15 and 30 days following randomization for evaluation of the occurrence of any trial endpoints or other adverse events.

Safety and efficacy will be based on data from randomized patients. An independent data and safety monitoring board (DSMB) will periodically review study results as well as the overall conduct of the study, and will make recommendations to the study Executive Steering Committee (ESC) to continue, stop or modify the study protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, at least 40 years of age, capable and willing to provide informed consent;
2. Patient must have received a diagnosis of COVID-19 infection within the last 24 hours;
3. Outpatient setting (not currently hospitalized or under immediate consideration for hospitalization);
4. Patient must possess at least one of the following high-risk criteria: 70 years or more of age, obesity (BMI ≥ 30 kg/m2), diabetes mellitus, uncontrolled hypertension (systolic blood pressure ≥150 mm Hg), known respiratory disease (including asthma or chronic obstructive pulmonary disease), known heart failure, known coronary disease, fever of ≥38.4°C within the last 48 hours, dyspnea at the time of presentation, bicytopenia, pancytopenia, or the combination of high neutrophil count and low lymphocyte count;
5. Female patient is either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile, or is of childbearing potential and practicing at least one method of contraception and preferably two complementary forms of contraception including a barrier method (e.g. male or female condoms, spermicides, sponges, foams, jellies, diaphragm, intrauterine device (IUD)) throughout the study and for 30 days after study completion;
6. Patient must be able and willing to comply with the requirements of this study protocol.

Exclusion Criteria:

1. Patient currently hospitalized or under immediate consideration for hospitalization;
2. Patient currently in shock or with hemodynamic instability;
3. Patient with inflammatory bowel disease (Crohn's disease or ulcerative colitis), chronic diarrhea or malabsorption;
4. Patient with pre-existent progressive neuromuscular disease;
5. Estimated Glomerular filtration rate (eGFR), using the MDRD equation for all subjects being considered for enrollment, with a cut-off of < 30 mL/m in/1.73m2;
6. Patient with a history of cirrhosis, chronic active hepatitis or severe hepatic disease;
7. Female patient who is pregnant, or breast-feeding or is considering becoming pregnant during the study or for 6 months after the last dose of study medication;
8. Patient currently taking colchicine for other indications (mainly chronic indications represented by Familial Mediterranean Fever or gout);
9. Patient with a history of an allergic reaction or significant sensitivity to colchicine;
10. Patient undergoing chemotherapy for cancer;
11. Patient is considered by the investigator, for any reason, to be an unsuitable candidate for the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4506 (Actual)
Dates: Start 2020-03-23 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude Tardif, MD, Principal Investigator — Montreal Heart Institute; Zohar Bassevitch, B.SC., Study Director — Montreal Health Innovations Coordinating Center
Locations (32):
- United States (16):
  - Mayo Clinic - Phoenix, Phoenix, Arizona
  - Yuma Regional Medical Center Cancer Center, Yuma, Arizona
  - Centric Health Resources Inc., Bakersfield, California
  - Westside Medical Associates of Los Angeles, Beverly Hills, California
  - Rancho Research Institute, Downey, California
  - University of California San Francisco - Zuckerberg San Francisco General Hospital, San Francisco, California
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - South Florida Research Organization, Medley, Florida
  - Miami Center for Advanced Cardiology, Miami Beach, Florida
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - North Mississippi Medical Clinics, Inc., Tupelo, Mississippi
  - New York Langone Health, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Baylor Scott & White Research Institute - Pharmacy, Dallas, Texas
  - University of Texas(UT) Southwestern Medical Center, Dallas, Texas
  - Spring Clinical Research, Houston, Texas
- Brazil (6):
  - Instituto do Coração (InCor), School of Medicine, University of Sao Paulo, São Paulo, São Paulo
  - Hospital Universitário Bragança Paulista, Bragança Paulista
  - Instituto Cruzaltense de Cardiologia, Cruz Alta
  - Hospital de Clínicas de Passo Fundo, Passo Fundo
  - Hospital de Clinicas de Porto Alegre, Porto Alegre
  - Hospital Samaritano Higienópolis, São Paulo
- Montreal Heart Institute, Montreal, Quebec, Canada
- Greece (2):
  - University General Hospital of Athens "Attikon", Chaïdári, Athens
  - General Hospital of Kozani "Mamatsio", Kozani
- Tread Research, Tygerberg Hospital, Cape Town, South Africa
- Spain (6):
  - Hospital Universitario La Paz, IdiPaz, La Paz, Madrid
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid

REFERENCES:
- [Derived] Alfehaid LS, Farah S, Omer A, Weber BN, Alkhezi O, Tawfik YMK, Shah AM, Libby P, Buckley LF. Drug-Drug Interactions and the Clinical Tolerability of Colchicine Among Patients With COVID-19: A Secondary Analysis of the COLCORONA Randomized Clinical Trial. JAMA Netw Open. 2024 Sep 3;7(9):e2431309. doi: 10.1001/jamanetworkopen.2024.31309. PMID 39240567
- [Derived] Mikolajewska A, Fischer AL, Piechotta V, Mueller A, Metzendorf MI, Becker M, Dorando E, Pacheco RL, Martimbianco ALC, Riera R, Skoetz N, Stegemann M. Colchicine for the treatment of COVID-19. Cochrane Database Syst Rev. 2021 Oct 18;10(10):CD015045. doi: 10.1002/14651858.CD015045. PMID 34658014
- [Derived] Tardif JC, Bouabdallaoui N, L'Allier PL, Gaudet D, Shah B, Pillinger MH, Lopez-Sendon J, da Luz P, Verret L, Audet S, Dupuis J, Denault A, Pelletier M, Tessier PA, Samson S, Fortin D, Tardif JD, Busseuil D, Goulet E, Lacoste C, Dubois A, Joshi AY, Waters DD, Hsue P, Lepor NE, Lesage F, Sainturet N, Roy-Clavel E, Bassevitch Z, Orfanos A, Stamatescu G, Gregoire JC, Busque L, Lavallee C, Hetu PO, Paquette JS, Deftereos SG, Levesque S, Cossette M, Nozza A, Chabot-Blanchet M, Dube MP, Guertin MC, Boivin G; COLCORONA Investigators. Colchicine for community-treated patients with COVID-19 (COLCORONA): a phase 3, randomised, double-blinded, adaptive, placebo-controlled, multicentre trial. Lancet Respir Med. 2021 Aug;9(8):924-932. doi: 10.1016/S2213-2600(21)00222-8. Epub 2021 May 27. PMID 34051877

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 18 patients were not included:
  * 11 study medication was not delivered at home;
  * 7 ineligible or condition deteriorated before study medication was delivered.
Groups:
- Placebo: Patients will receive the placebo 0.5 mg per os (PO) twice daily for the first 3 days and then once daily for the last 27 days. If a dose is missed, it should not be replaced.
Period: Overall Study
Arm/Group | Colchicine | Placebo
Started | 2235 | 2253
Completed | 2192 | 2189
Not Completed | 43 | 64
Not completed — Withdrawal by Subject | 33 | 47
Not completed — Death | 5 | 9
Not completed — Lost to Follow-up | 4 | 8
Not completed — Admitted to Hospital and Intubated | 1 | 0

BASELINE CHARACTERISTICS:
Population: Characteristics of the patients at randomisation in the intent-to-treat population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Colchicine | Placebo | Total
Number analyzed (Participants) | 2235 | 2253 | 4488
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53.0 [47.0 to 61.0] | 54.0 [47.0 to 61.0] | 54.0 [47.0 to 61.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1238 | 1183 | 2421
  Male | 997 | 1070 | 2067
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 327 | 349 | 676
  Not Hispanic or Latino | 1869 | 1872 | 3741
  Unknown or Not Reported | 39 | 32 | 71
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 9 | 14
  Asian | 23 | 20 | 43
  Native Hawaiian or Other Pacific Islander | 7 | 7 | 14
  Black or African American | 114 | 116 | 230
  White | 2084 | 2092 | 4176
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 0 | 5 | 5
Region of Enrollment [Number; unit: participants]
  Canada | 1817 | 1830 | 3647
  United States | 244 | 244 | 488
  South Africa | 0 | 2 | 2
  Spain | 94 | 94 | 188
  Brazil | 79 | 82 | 161
  Greece | 1 | 1 | 2
History of Respiratory Disease [Count of Participants; unit: Participants]
  Yes | 583 | 605 | 1188
  No | 1652 | 1647 | 3299
  Not Reported | 0 | 1 | 1
History of Diabetes [Count of Participants; unit: Participants]
  Yes | 444 | 450 | 894
  No | 1791 | 1803 | 3594
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.0 (6.2) | 30.0 (6.3) | 30.0 (6.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Died or Were Hospitalized Due to COVID-19 Infection in the 30 Days Following Randomization.
Description: The primary endpoint will be the composite of death or hospitalization due to COVID-19 infection in the 30 days following randomization.
Time Frame: 30 days post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine | Placebo
Number analyzed (Participants) | 2235 | 2253
Participants | 104 | 131
Statistical Analysis 1: Comparison: Colchicine vs Placebo; Test type: Superiority; p = 0.081, Chi-squared; Odds Ratio (OR) = 0.79, 95.1% CI 2-sided [0.61 to 1.03]

2. Secondary Outcome: Number of Deaths in the 30 Days Following Randomization.
Description: The secondary endpoint consisted of two components of the composite primary endpoint and included death in the 30 days following randomization.
Time Frame: 30 days post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine | Placebo
Number analyzed (Participants) | 2235 | 2253
Participants | 5 | 9
Statistical Analysis 1: Comparison: Colchicine vs Placebo; Test type: Superiority; p = 0.291, Chi-squared; Odds Ratio (OR) = 0.56, 95% CI 2-sided [0.19 to 1.67]

3. Secondary Outcome: Number of Participants Who Were Hospitalized Due to COVID-19 Infection in the 30 Days Following Randomization.
Description: The secondary endpoint consisted of two components of the composite primary endpoint and included hospitalization due to COVID-19 infection in the 30 days following randomization.
Time Frame: 30 days post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine | Placebo
Number analyzed (Participants) | 2235 | 2253
Participants | 101 | 128
Statistical Analysis 1: Comparison: Colchicine vs Placebo; Test type: Superiority; p = 0.077, Chi-squared; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.60 to 1.03]

4. Secondary Outcome: Number of Participants Who Required Mechanical Ventilation in the 30 Days Following Randomization.
Description: The secondary endpoint is the need for mechanical ventilation in the 30 days following randomization.
Time Frame: 30 days post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine | Placebo
Number analyzed (Participants) | 2235 | 2253
Participants | 11 | 21
Statistical Analysis 1: Comparison: Colchicine vs Placebo; Test type: Superiority; p = 0.080, Chi-squared; Odds Ratio (OR) = 0.53, 95% CI 2-sided [0.25 to 1.09]

5. Other Pre Specified Outcome: Number of Participants Who Died or Were Hospitalized Due to COVID-19 Infection in the 30 Days Following Randomization in the Subgroup of Patients With PCR-confirmed COVID-19.
Description: In the prespecified analysis of the 4159 patients with Covid-19 confirmed by PCR, the primary endpoint (composite of death or hospitalization due to Covid-19 infection in the 30 Days following randomization) was compared between the two treatment groups.
Time Frame: 30 Days post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine | Placebo
Number analyzed (Participants) | 2075 | 2084
Participants | 96 | 126
Statistical Analysis 1: Comparison: Colchicine vs Placebo; Test type: Superiority; p = 0.042, Regression, Logistic — P-Value is for the comparison of the treatment group within patients with Covid-19 confirmed by PCR; Logistic-regression model including the treatment group, the PCR-confirmed Covid-19 subgroup factor (yes/no) and their interaction was performed; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.57 to 0.99]

6. Other Pre Specified Outcome: Number of Participants Who Died or Were Hospitalized Due to COVID-19 Infection in the 30 Days Following Randomization by Sex
Description: NIH-required analysis. The primary endpoint will be the composite of death or hospitalization due to COVID-19 infection in the 30 days following randomization by Sex.
Time Frame: 30 Days post randomization
Population: Data were stratified by sex.
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine | Placebo
Number analyzed (Participants) | 2235 | 2253
Participants
  Male: number analyzed (Participants) | 997 | 1070
  Male | 58 | 90
  Female: number analyzed (Participants) | 1238 | 1183
  Female | 46 | 41

7. Other Pre Specified Outcome: Number of Participants Who Died or Were Hospitalized Due to COVID-19 Infection in the 30 Days Following Randomization by Race
Description: NIH-required analysis. The primary endpoint will be the composite of death or hospitalization due to COVID-19 infection in the 30 days following randomization by Race.
Time Frame: 30 Days post randomization
Population: Data were stratified by race.
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine | Placebo
Number analyzed (Participants) | 2235 | 2253
Participants
  American Indian or Alaska Native: number analyzed (Participants) | 5 | 9
  American Indian or Alaska Native | 1 | 2
  Asian: number analyzed (Participants) | 23 | 20
  Asian | 1 | 3
  Black: number analyzed (Participants) | 114 | 116
  Black | 3 | 6
  Native Hawaiian or other Pacific Islander: number analyzed (Participants) | 7 | 7
  Native Hawaiian or other Pacific Islander | 1 | 0
  White: number analyzed (Participants) | 2084 | 2092
  White | 98 | 120
  More than one race: number analyzed (Participants) | 2 | 4
  More than one race | 0 | 0
  Not reported or unknown: number analyzed (Participants) | 0 | 5
  Not reported or unknown | 0 | 0

8. Other Pre Specified Outcome: Number of Participants Who Died or Were Hospitalized Due to COVID-19 Infection in the 30 Days Following Randomization by Ethnicity.
Description: NIH-required analysis. The primary endpoint will be the composite of death or hospitalization due to COVID-19 infection in the 30 days following randomization by Ethnicity.
Time Frame: 30 Days post randomization
Population: Data were stratified by ethnicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine | Placebo
Number analyzed (Participants) | 2235 | 2253
Participants
  Hispanic or Latino: number analyzed (Participants) | 327 | 349
  Hispanic or Latino | 20 | 24
  Not Hispanic or Latino: number analyzed (Participants) | 1869 | 1872
  Not Hispanic or Latino | 82 | 106
  Not reported or unknown: number analyzed (Participants) | 39 | 32
  Not reported or unknown | 2 | 1

ADVERSE EVENTS:
Time Frame: From randomization/baseline to End of Study visit which planned 30 days after baseline.
Description: 2 additional Serious Adverse Events were added to the definition :
  * cancer;
  * overdose (intentional or accidental).
  Adverse events reporting are presented on the Safety population where subjects took at least one dose of study medication and are assigned according to the true treatment received.
  The Safety population includes 2217 subjects have received placebo and 2195 subjects have received colchicine.
Arm/Group | Colchicine | Placebo
All-Cause Mortality (participants affected / at risk) | 5/2195 | 9/2217
Serious Adverse Events (participants affected / at risk) | 108/2195 | 139/2217
Other Adverse Events (participants affected / at risk) | 524/2195 | 328/2217
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Colchicine (N=2195) | Placebo (N=2217)
Arrhythmia (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Death (General disorders) | 1 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Blood magnesium abnormal (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 6
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 2
Tachycardia (Cardiac disorders) | 2 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 3 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Corona virus infection (Infections and infestations) | 2 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 63 | 92
Pneumonia bacterial (Infections and infestations) | 4 | 2
Pneumonia viral (Infections and infestations) | 2 | 2
Pyelonephritis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 2
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 3
Loss of proprioception (Nervous system disorders) | 0 | 1
Multiple sclerosis (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 11 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 12 | 13
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Colchicine (N=2195) | Placebo (N=2217)
Abdominal discomfort (Gastrointestinal disorders) | 7 | 3
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 28 | 18
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 7
Diarrhoea (Gastrointestinal disorders) | 300 | 161
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 8 | 13
Epigastric discomfort (Gastrointestinal disorders) | 1 | 2
Faeces soft (Gastrointestinal disorders) | 10 | 2
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastric disorder (Gastrointestinal disorders) | 12 | 8
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 114 | 72
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 43 | 47
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 6 | 4

LIMITATIONS AND CAVEATS:
Due to several considerations (logistical, human and budgetary), the study was stopped early. Furthermore, stopping the study after approximately 4500 patients had completed their 30-day follow-up would allow to communicate results in January 2021 in the hope of preventing complications of COVID-19 in ambulatory patients, instead of delivering results anywhere between April and October 2021 at a time when vaccination efforts might be successful.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/82/NCT04322682/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-25): https://cdn.clinicaltrials.gov/large-docs/82/NCT04322682/SAP_001.pdf